CLINICAL TRIAL: NCT04035421
Title: Diet, Physical Activity, and Sleep Habits
Acronym: DPAS
Status: Completed | Type: Observational
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Other Study IDs: UTK IRB-19-05178-XP
Record Dates: First submitted 2019-07-13; First posted 2019-07-29 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Diet Habit
Keywords: Social Rhythm Metric; Chronotype; Young adult
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to observe if consistency in a young adult's schedule is related to health factors and outcomes, such as diet quality, amount of physical activity and sleep, and weight.

DETAILED DESCRIPTION:
During young adulthood, patterns regarding physical activity,1,2 dietary intake,3 and weight status4 are established that track into later life and can impact health. Social and physical cues also impact patterns-particularly those cues that may influence biological and behavioral rhythms which can influence the Circadian Timing System (CTS).5 Chronotype, the timing of sleep patterns, is closely tied to the CTS as it reflects sleep in relation to the light and dark cycle, with morning-type (MT) having a pattern that should assist with better entrainment (sleep better entrained to the physical cues of light/dark).6 Research has found that chronotype is related to several areas important to health, including diet,6-11 physical activity,12-14 weight regulation.15-18. As a whole, research in this area suggests that MT individuals are more likely to consume a healthier eating pattern, be more physically active, and more successfully manage their weight. However, the research in this area for young adults is limited.

While there has been research regarding chronotype and diet, activity, and weight management, there is a paucity of research on the relationship between social cues and social rhythms, which also influence the CTS, and health related outcomes. Social rhythms, as measured by the Social Rhythm Metric (SRM), are related to chronotype, such that MT is related to a higher SRM.19-21 Due to the relationship between SRM and chronotype, and chronotype and diet, physical activity, and weight management, it would be anticipated that SRM is also related to these health outcomes. Specifically, it would be anticipated that more consistent social rhythms (higher SRM) would be related to a healthier eating pattern, greater physical activity, and weight management. However, this relationship has never been investigated.

Therefore, to better understand how social rhythms, which are triggered by social cues, are related to health, this investigation will be assessing both chronotype and SRM and collecting measures on diet quality, via food records, physical activity and sleep, via accelerometers, and anthropometrics, via BMI. The population of interest for this study is specifically young adults because young adulthood is a time period when health patterns are established for the rest of life. This study aims to observe if consistency in a young adult's schedule is related to health factors and outcomes, such as diet quality, amount of physical activity and sleep, and weight.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-35 years
* Able to pass the Physical Activity Readiness Questionnaire for Everyone (PAR-Q+) indicating that they have no health conditions that limit their ability to engage in physical activity
* Access to an email address and internet each day during their participation
* An town when all measures are collected
* Taking classes and/or working a job when all measures are collected

Exclusion Criteria:

* Pregnant
* Allergy to stainless steel, making the participant unable to wear Body Media Armband
* Dietary restrictions of any kind
* Shift work, here defined as having to work a shift for any period of time between the hours of 12 am and 6 am

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young adult between the ages of 18 and 35 years, taking classes and/or working, able to engage in physical activity, and having no dietary restrictions.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2019-07-13 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Diet Quality 1 | Through study completion, 1 week
  Healthy Eating Index Score calculated using a three-day food record
Diet Quality 2 | Through study completion, 1 week
  Total energy intake will be assessed using a three-day food record
Physical Activity 1 | Through study completion, 1 week
  Minutes of moderate to vigorous physical activity will be assessed using SenseWear Armbands
Physical Activity 2 | Through study completion, 1 week
  Energy expenditure from moderate to vigorous physical activity will be assessed using SenseWear Armbands
Sleep 1 | Through study completion, 1 week
  Length of sleep will be assessed using SenseWear Armbands
Sleep 2 | Through study completion, 1 week
  Sleep efficiency will be assessed using SenseWear Armbands

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Baseline appointment
  BMI will be calculated using height and weight measurements
Body Composition | Baseline appointment
  Body fat percentage will be assessed using the Body Composition Analyzer TBF-300 (TANITA Corporation, Tokyo, Japan)
Chronotype | Baseline appointment
  Chronotype will be assessed using the Composite Score for Morningness

CONTACTS AND LOCATIONS:
Overall Officials: Hollie Raynor, PhD, Principal Investigator — University of Tennessee Knoxville
Locations (1):
- Healthy Eating and Activity Lab, University of Tennessee, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caspersen CJ, Pereira MA, Curran KM. Changes in physical activity patterns in the United States, by sex and cross-sectional age. Med Sci Sports Exerc. 2000 Sep;32(9):1601-9. doi: 10.1097/00005768-200009000-00013. PMID 10994912
- [Background] Nelson MC, Story M, Larson NI, Neumark-Sztainer D, Lytle LA. Emerging adulthood and college-aged youth: an overlooked age for weight-related behavior change. Obesity (Silver Spring). 2008 Oct;16(10):2205-11. doi: 10.1038/oby.2008.365. No abstract available. PMID 18719665
- [Background] Dunn JE, Liu K, Greenland P, Hilner JE, Jacobs DR Jr. Seven-year tracking of dietary factors in young adults: the CARDIA study. Am J Prev Med. 2000 Jan;18(1):38-45. doi: 10.1016/s0749-3797(99)00114-2. PMID 10808981
- [Background] Serdula MK, Ivery D, Coates RJ, Freedman DS, Williamson DF, Byers T. Do obese children become obese adults? A review of the literature. Prev Med. 1993 Mar;22(2):167-77. doi: 10.1006/pmed.1993.1014. PMID 8483856
- [Background] Monk TH, Flaherty JF, Frank E, Hoskinson K, Kupfer DJ. The Social Rhythm Metric. An instrument to quantify the daily rhythms of life. J Nerv Ment Dis. 1990 Feb;178(2):120-6. doi: 10.1097/00005053-199002000-00007. PMID 2299336
- [Background] Wright KP Jr, McHill AW, Birks BR, Griffin BR, Rusterholz T, Chinoy ED. Entrainment of the human circadian clock to the natural light-dark cycle. Curr Biol. 2013 Aug 19;23(16):1554-8. doi: 10.1016/j.cub.2013.06.039. Epub 2013 Aug 1. PMID 23910656
- [Background] Fleig D, Randler C. Association between chronotype and diet in adolescents based on food logs. Eat Behav. 2009 Apr;10(2):115-8. doi: 10.1016/j.eatbeh.2009.03.002. Epub 2009 Mar 29. PMID 19447353
- [Background] Gontijo CA, Cabral BBM, Balieiro LCT, Teixeira GP, Fahmy WM, Maia YCP, Crispim CA. Time-related eating patterns and chronotype are associated with diet quality in pregnant women. Chronobiol Int. 2019 Jan;36(1):75-84. doi: 10.1080/07420528.2018.1518328. Epub 2018 Sep 13. PMID 30212228
- [Background] Kogevinas M, Espinosa A, Castello A, Gomez-Acebo I, Guevara M, Martin V, Amiano P, Alguacil J, Peiro R, Moreno V, Costas L, Fernandez-Tardon G, Jimenez JJ, Marcos-Gragera R, Perez-Gomez B, Llorca J, Moreno-Iribas C, Fernandez-Villa T, Oribe M, Aragones N, Papantoniou K, Pollan M, Castano-Vinyals G, Romaguera D. Effect of mistimed eating patterns on breast and prostate cancer risk (MCC-Spain Study). Int J Cancer. 2018 Nov 15;143(10):2380-2389. doi: 10.1002/ijc.31649. Epub 2018 Jul 17. PMID 30016830
- [Background] Maukonen M, Kanerva N, Partonen T, Mannisto S. Chronotype and energy intake timing in relation to changes in anthropometrics: a 7-year follow-up study in adults. Chronobiol Int. 2019 Jan;36(1):27-41. doi: 10.1080/07420528.2018.1515772. Epub 2018 Sep 13. PMID 30212231
- [Background] Rossbach S, Diederichs T, Nothlings U, Buyken AE, Alexy U. Relevance of chronotype for eating patterns in adolescents. Chronobiol Int. 2018 Mar;35(3):336-347. doi: 10.1080/07420528.2017.1406493. Epub 2017 Dec 12. PMID 29231764
- [Background] Harrex HAL, Skeaff SA, Black KE, Davison BK, Haszard JJ, Meredith-Jones K, Quigg R, Saeedi P, Stoner L, Wong JE, Skidmore PML. Sleep timing is associated with diet and physical activity levels in 9-11-year-old children from Dunedin, New Zealand: the PEDALS study. J Sleep Res. 2018 Aug;27(4):e12634. doi: 10.1111/jsr.12634. Epub 2017 Nov 20. PMID 29160021
- [Background] Olds TS, Maher CA, Matricciani L. Sleep duration or bedtime? Exploring the relationship between sleep habits and weight status and activity patterns. Sleep. 2011 Oct 1;34(10):1299-307. doi: 10.5665/SLEEP.1266. PMID 21966061
- [Background] Shechter A, St-Onge MP. Delayed sleep timing is associated with low levels of free-living physical activity in normal sleeping adults. Sleep Med. 2014 Dec;15(12):1586-9. doi: 10.1016/j.sleep.2014.07.010. Epub 2014 Sep 2. PMID 25311835
- [Background] Arora T, Taheri S. Associations among late chronotype, body mass index and dietary behaviors in young adolescents. Int J Obes (Lond). 2015 Jan;39(1):39-44. doi: 10.1038/ijo.2014.157. Epub 2014 Aug 19. PMID 25135376
- [Background] Culnan E, Kloss JD, Grandner M. A prospective study of weight gain associated with chronotype among college freshmen. Chronobiol Int. 2013 Jun;30(5):682-90. doi: 10.3109/07420528.2013.782311. Epub 2013 May 20. PMID 23688114
- [Background] Ross KM, Graham Thomas J, Wing RR. Successful weight loss maintenance associated with morning chronotype and better sleep quality. J Behav Med. 2016 Jun;39(3):465-71. doi: 10.1007/s10865-015-9704-8. Epub 2015 Dec 10. PMID 26660638
- [Background] Ruiz-Lozano T, Vidal J, de Hollanda A, Scheer FAJL, Garaulet M, Izquierdo-Pulido M. Timing of food intake is associated with weight loss evolution in severe obese patients after bariatric surgery. Clin Nutr. 2016 Dec;35(6):1308-1314. doi: 10.1016/j.clnu.2016.02.007. Epub 2016 Feb 16. PMID 26948400
- [Background] Martin JS, Hebert M, Ledoux E, Gaudreault M, Laberge L. Relationship of chronotype to sleep, light exposure, and work-related fatigue in student workers. Chronobiol Int. 2012 Apr;29(3):295-304. doi: 10.3109/07420528.2011.653656. PMID 22390242
- [Background] Mongrain V, Carrier J, Dumont M. Chronotype and sex effects on sleep architecture and quantitative sleep EEG in healthy young adults. Sleep. 2005 Jul;28(7):819-27. doi: 10.1093/sleep/28.7.819. PMID 16124660
- [Background] Monk TH, Buysse DJ, Potts JM, DeGrazia JM, Kupfer DJ. Morningness-eveningness and lifestyle regularity. Chronobiol Int. 2004 May;21(3):435-43. doi: 10.1081/cbi-120038614. PMID 15332448

DOCUMENTS (1):
  • Informed Consent Form (2019-07-23): https://cdn.clinicaltrials.gov/large-docs/21/NCT04035421/ICF_000.pdf